CLINICAL TRIAL: NCT04094181
Title: VPRIV® Non-Interventional Study in Patients Previously Treated With Other Enzyme Replacement Therapies (ERTs)/Substrate Reduction Therapies (SRTs)
Brief Title: A Study of VPRIV in Participants With Gaucher Disease Previously Treated With Other Enzyme Replacement Therapies or Substrate Reduction Therapies
Status: Terminated | Type: Observational
Why Stopped: The decision was taken after careful consideration relating to recruitment challenges that could impact the scientific value of the study.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP669-405; EUPAS42338 (Registry Identifier: EUPAS)
Record Dates: First submitted 2019-09-17; First posted 2019-09-18 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VPRIV Participants: Participants who has been transitioned from ERTs/SRTs to VPRIV, the data will be collected retrospectively from time of transition until the point at which participant begins in this study and then will be followed up prospectively for 12 months.

SUMMARY:
The main aim of this study is to describe the safety profile of velaglucerase alfa (VPRIV) in participants with Gaucher disease type 1. Participants will be transitioning from other enzyme replacement therapies or substrate reduction therapies to VPRIV. Some participants may have already transitioned to treatment with VPRIV before this study started.

In this study, data on VPRIV will be collected from the medical records of participants who already transitioned to VPRIV before this study started. Other participants will join this study when they transition to VPRIV. All participants will be followed to allow for 12 months of observation from time of transition to VPRIV.

The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant with GD1 currently being treated with an ERT/SRT other than VPRIV for at least 6 months before baseline enrolment; or participant previously treated with another ERT/ SRT for at least 6 months prior to transitioning to VPRIV..
* Participant or legally authorized representative has provided written informed consent.

Exclusion Criteria:

* In the opinion of the investigator, participant is at high risk of non-compliance.
* In the opinion of the investigator, participant is unsuitable in any other way to participate in this study.
* Participant is pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants included in the study will have a diagnosis of Type 1 GD and be in enzyme/substrate replacement therapy other than VPRIV, for at least 6 months prior to enrolment in the study, or have been previously treated with an ERT/SRT other than VPRIV for a minimum of 6 months prior to transitioning to VPRIV.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) Following the Transition From Other ERTs/SRTs to VPRIV | Baseline up to 12 months
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Number of participants transitioning from other ERTs/SRTs to VPRIV with AEs will be reported.

SECONDARY OUTCOMES:
Change From Baseline in Use of Glucosylspingosine (Lyso-Gb1) Biomarker | Baseline, Month 12
  Change in use of Lyso-Gb1 by participants following the transition from other ERTs/SRTs to velaglucerase alfa (VPRIV) will be assessed.
Change From Baseline in Gaucher Disease Questionnaire Patient Reported Outcomes (PRO) Score at Month 12 | Baseline, Month 12
  Gaucher disease questionnaire (PRO) scores will be calculated for each adult participant. The questionnaire asks how much the participant is affected by the Gaucher disease. A total summated score is calculated and ranges from 0 to 100 with higher scores indicating more severe impairment and worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- University of Alberta/Medical Genetics Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe84db2bf003ab47b16